CLINICAL TRIAL: NCT03596606
Title: Additional Effects of Therapeutic Exercises Under a Behavioral Umbrella for Chronic Temporomandibular Disorders Treatment. A Double-blind Randomized Clinical Trial
Brief Title: Additional Effects of Therapeutic Exercises Under a Behavioral Umbrella for Chronic Temporomandibular Disorders Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maxilofacial Institute Bara Gaseni (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2018/33-CMF-HUSC
Record Dates: First submitted 2018-06-28; First posted 2018-07-24 (Actual); Last update posted 2023-06-02 (Actual); Status verified 2023-05

CONDITIONS: Temporomandibular Joint Dysfunction Syndrome
Keywords: Chronic Facial Pain; Osteopathic Manual treatment; Therapeutic Exercise
MeSH Terms: conditions — Temporomandibular Joint Dysfunction Syndrome

STUDY DESIGN:
Intervention Model Description: Both groups will be treated with Osteopathic Treatment and in one of them it will be added the intervention with cognition targeted myofunctional motor control exercises.
Who Masked: Investigator
Masking Description: The principal evaluator will be blinded in relation to the study groups. The person responsible for taking the variables (baseline data, reassessments and data analysis) will be a therapist and a medical doctor unrelated to the recruitment and treatment. Due to the nature of the interventions, it is not possible to mask the therapist responsible for the interventions.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Myofunctional Motor Control Exercises (Experimental): Both groups will be treated with Manual treatment and in one of them the myofunctional motor control treatment will be added as intervention. The experimental group will be the one that will receive the combined treatment.
  The patient will receive five sessions, one session every week.
  Interventions: Procedure: Manual Treatment; Procedure: Myofunctional Motor control exercises
- Manual Treatment (Active Comparator): The control group will receive only Manual treatment (TO). The patient will receive five sessions, one session every week.
  Interventions: Procedure: Manual Treatment

INTERVENTIONS:
Procedure: Manual Treatment — The manual treatment will be adapted to each patient at the discretion of the therapist, being able to select all or part of the following osteopathic techniques in each session.
  * Soft tissue techniques.
  * Articulatory techniques applied at cervical level
  * Osteopathic manipulation techniques applied at the affected jaw/s.
  * Functional Indirect technique at the level of the affected jaw/s: For Type I or II diagnosis.
Procedure: Myofunctional Motor control exercises — The protocol is a set of 8 exercises to improve the execution of the function in the stomatognathic and cervical area.
  The therapist explains the objectives of the exercises and the patient performs it after each session and at home three times a day.
  The first day before performing the myofunctional exercises, will be an explanatory talk prior to the exercises in order to educate the patient. The second day, before doing the exercises, will review the concept of memory of pain and the benefits of doing the exercises
  Arms: Myofunctional Motor Control Exercises

SUMMARY:
Temporomandibular dysfunction (TMD) It's one of the main causes of oro-facial chronic pain. The psychological aspects of patients with TMD have a huge importance, affecting their ability to manage pain and interfering with the resolution of the picture.

Different studies analyse Manual therapy (MT) and motor control exercises (MC) as a whole or separately. In these cases, MT with MC shows promising results. Despite this, MC do not suggest adding significant improvement at least at short term. In the other side, according to a recent research line, MC with education is the clue for chronic pain management. This leads us to think that it should be studied more carefully if MC performed with a cognitive approach adds beneficial effect to MT not only in purely mechanical aspects but also in psycho-social aspects of the individual and at longer term.

HYPOTHESIS The combination of MT and MC is more effective than MT applied in a unique way for the treatment of pain, function and psycho-social symptoms associated with chronic TMD.

DETAILED DESCRIPTION:
TMD is an alteration of the jaw function associated with disorders at the mastication muscles, mandibular joint and its associated tissues. It constitutes a major health problem since it's one of the main causes of oro-facial chronic pain and interferes with daily life. It is associated with headache, otological symptoms, cervical dysfunction and alterations in posture at the cervical level. The TMD involves genetic, anatomical, hormonal factors, traumatisms, motor behaviour, psycho-social aspects and occlusal problems.

The psychological aspects of patients with TMD have a huge importance, affecting their ability to manage pain and interfering with the resolution of the picture. It can even cause the pain to become chronic. The most prevalent symptoms in TMD are somatization and depression. Chronic pain can lead to plastic changes in the brain that lead to hyper-excitability of the central nervous system. Persistent pain produces protective memories that involve antalgic behaviour, avoidance and kinesiophobia. The literature shows that somatization, depression, fear of pain, fear of movement and catastrophism in conjunction with the amplification of pain are key factors in the chronification of TMD.

The TMD treatment must provide the ideal circumstances for the repair and adaptation. The TMD is usually a benign self-limiting process, so the guidelines always recommend non-invasive, reversible treatments in the first instance and within the bio-psycho-social approach.

For conservative management, the most evidence-based approach is manual therapy (MT). The one that has demonstrated more effectiveness is the mobilisation with impulse and / or mobilisation both at cervical and mandibular level. MT improves motor response, range of motion and modulates pain intensity via peripheral, medullary and supraspinal mechanisms. Theories suggest that hypoalgesia is caused by several mechanisms mediated by the periaqueductal gray substance.

Different studies analyse MT and motor control exercises (MC) as a whole or separately, comparing them with other therapies such as education, splints, medication, botulinum toxin, arthroplasty and arthroscopy. In these cases, MT with MC are superior to these therapies. Despite this, MC exercises do not suggest adding significant improvement in the treatment of TMD, at least in the short term. Shafer et al., In a recent systematic review, state that there is currently no evidence for the use of MC exercises of any kind for the management of TMD in general. However, according to a recent research line MC with education is the clue for the management of chronic pain. The objective of the exercises is to perform a cognitive approach to provide the desensitization of the central nervous system, generate new memories and eliminate the protective movement associated with chronic pain. It also promotes eliminating catastrophism, avoidance and fear of pain behaviour associated with chronification. This leads us to think that it should be studied more carefully if CM performed with a cognitive approach adds beneficial effect to MT in the treatment of chronic TMD not only in purely mechanical aspects but also in psycho social aspects of the individual and longer term.

The current studies are of low quality, have biases in the selection, randomisation and allocation concealment. Patient selection and diagnostic criteria are not standardised. There is a lack of blind of the evaluator and examiner. The therapy or exercise is not well described making them difficult to reproduce. The new lines of research require more detail about the type of exercise to be performed and the MT applied as recommended by the intervention report guides.

HYPOTHESIS The combination of MT and Myofunctional MC (MMC) is more effective than MT applied in a unique way for the treatment of pain, function and psycho social symptoms associated with chronic TMD.

ELIGIBILITY:
Inclusion Criteria:

* Primary diagnosis of TMD type: I myofascial and or II displacement of disc and or III other arthralgias. According to the diagnostic criteria of Dworkin S. Et al. The clinical examination and algorithms that will be carried are the ones included in the the axis I of the Diagnostic criteria for TMD (DC/TMD). We will use the Spanish version.
* 6 months of TMD evolution and pain in the last 30 days.
* Signs of pain and disability of at least 7 points on the CF-PDI.
* Normal neurological examination.
* Normal orthopantomography (without fracture or severe joint bone disease).
* To accept the participation and sign the informed consent.

Exclusion Criteria:

* Severe dermatological or intrabuccal problems, head or neck injuries.
* Orthopantomography with recent fractures or severe articular bone pathology.
* Previous treatment (three months before) with manual therapy splints or acupuncture.
* Previous diagnosis of severe psychiatric disorder.
* Systemic, rheumatologic or neurodegenerative diseases.
* Previous diagnosis of primary headache or unilateral neck pain of recent appearance.
* Associated clinic of neurological pain, radiculopathy or myelopathy.
* Not understanding Castilian or Catalan.

Ages: 5 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2019-09-16 (Actual); Primary Completion 2023-01-28 (Actual); Study Completion 2023-01-28 (Actual)

PRIMARY OUTCOMES:
Change from Baseline Cranio Facial Pain and Disability Index during 3 months (CF-PDI) | 5 measures: Before the first intervention (CF-PDI1_ baseline data), 2 weeks later after the second session (CF-PDI2), 5 weeks later after the last session (CF-PDI3), 7 weeks later (CF-PDI4) and up to 3 months (CF-PDI5).
  It contains 21 Items divided into two sub-scales. The first sub-scale measures pain and associated disability. The second sub-scale measures the functional status of the jaw. The questionnaire scores from 0 to 63 points and the relevant minimum change is 7 points.

SECONDARY OUTCOMES:
Change from Baseline Mandibular Opening without pain during 3 months (MO) | 5 measures: Before the first intervention (MO1_ baseline data), 2 weeks later after the second session (MO2), 5 weeks later after the last session (MO3), 7 weeks later (MO4) and up to 3 months (MO5).
  It will be measured with a vernier caliper with an accuracy of 0.5 millimeters. The distance between the upper and lower central incisors will be measured. The measure will be taken with the patient sitting on the assessor's chair. It is considered a clinically relevant improvement an opening difference of 6mm.
Change from Baseline Position of the head during 3 months (CROM) | 5 measures: Before the first intervention (CROM1_ baseline data), 2 weeks later after the second session (CROM2), 5 weeks later after the last session (CROM3), 7 weeks later (CROM4) and up to 3 months (CROM5).
  The position of the head measured with the "Cervical Range of Motion "(CROM). The minimum relevant change is considered 1.27 cm.
Change from Baseline Occlusal force distribution during 3 months (FD) | 5 measures: Before the first intervention (FD1_ baseline data), 2 weeks later after the second session (FD2), 5 weeks later after the last session (FD3), 7 weeks later (FD4) and up to 3 months (FD5).
  It will be measured with the Occlusal T-Scan ® analysis system (Teskcan Inc., South Boston, MA, USA) that records different parameters of the dynamics of bite. Uses a thin and reusable intraoral sensor in the form of an arch dental. Obtains quantitative values of the bite.
  The value of the force of the bite is expressed:
  • In relation to the forces of the left side and the forces of the right side. The perfect balance would be 1. It will be the lateral ratio distribution.
Change from Baseline Pain Catastrophism scale during 3 months (PCS) | 5 measures: Before the first intervention (PCS1_ baseline data), 2 weeks later after the second session (PCS2), 5 weeks later after the last session (PCS3), 7 weeks later (PCS4) and up to 3 months (PCS5).
  It consists of 3 subscales (impotence, rumination and magnification). The minimum relevant change is identified in 9.1 points.
Change from Baseline Kinesiophobia during 3 months (TSK-11) | 5 measures: Before the first intervention (TSK1_ baseline data), 2 weeks later after the second session (TSK2), 5 weeks later after the last session (TSK3), 7 weeks later (TSK4) and up to 3 months (TSK5).
  The Spanish version TSK-11 is a self-assessment tool that evaluates the fear of reinjury due to movement. The score goes from 11 to 44 points. Higher results indicate high values of fear of movement, pain and injury itself. The minimum relevant change is 5,659.

CONTACTS AND LOCATIONS:
Overall Officials: Cristian Justribo manion, MSc, Principal Investigator
Locations (1):
- Calle Londres, 28, 4, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Armijo-Olivo S, Pitance L, Singh V, Neto F, Thie N, Michelotti A. Effectiveness of Manual Therapy and Therapeutic Exercise for Temporomandibular Disorders: Systematic Review and Meta-Analysis. Phys Ther. 2016 Jan;96(1):9-25. doi: 10.2522/ptj.20140548. Epub 2015 Aug 20. PMID 26294683
- [Background] Chaves TC, Turci AM, Pinheiro CF, Sousa LM, Grossi DB. Static body postural misalignment in individuals with temporomandibular disorders: a systematic review. Braz J Phys Ther. 2014 Nov-Dec;18(6):481-501. doi: 10.1590/bjpt-rbf.2014.0061. Epub 2014 Oct 31. PMID 25590441
- [Background] Butts R, Dunning J, Perreault T, Mettille J, Escaloni J. Pathoanatomical characteristics of temporomandibular dysfunction: Where do we stand? (Narrative review part 1). J Bodyw Mov Ther. 2017 Jul;21(3):534-540. doi: 10.1016/j.jbmt.2017.05.017. Epub 2017 May 31. PMID 28750961
- [Background] Celic R, Panduric J, Dulcic N. Psychologic status in patients with temporomandibular disorders. Int J Prosthodont. 2006 Jan-Feb;19(1):28-9. PMID 16479755
- [Background] Nijs J, Lluch Girbes E, Lundberg M, Malfliet A, Sterling M. Exercise therapy for chronic musculoskeletal pain: Innovation by altering pain memories. Man Ther. 2015 Feb;20(1):216-20. doi: 10.1016/j.math.2014.07.004. Epub 2014 Jul 18. PMID 25090974
- [Background] Maisa Soares G, Rizzatti-Barbosa CM. Chronicity factors of temporomandibular disorders: a critical review of the literature. Braz Oral Res. 2015;29:S1806-83242015000100300. doi: 10.1590/1807-3107BOR-2015.vol29.0018. Epub 2015 Jan 13. PMID 25590505
- [Background] Butts R, Dunning J, Pavkovich R, Mettille J, Mourad F. Conservative management of temporomandibular dysfunction: A literature review with implications for clinical practice guidelines (Narrative review part 2). J Bodyw Mov Ther. 2017 Jul;21(3):541-548. doi: 10.1016/j.jbmt.2017.05.021. Epub 2017 Jun 1. PMID 28750962
- [Background] Martins WR, Blasczyk JC, Aparecida Furlan de Oliveira M, Lagoa Goncalves KF, Bonini-Rocha AC, Dugailly PM, de Oliveira RJ. Efficacy of musculoskeletal manual approach in the treatment of temporomandibular joint disorder: A systematic review with meta-analysis. Man Ther. 2016 Feb;21:10-7. doi: 10.1016/j.math.2015.06.009. Epub 2015 Jun 25. PMID 26144684
- [Background] Monaco A, Cozzolino V, Cattaneo R, Cutilli T, Spadaro A. Osteopathic manipulative treatment (OMT) effects on mandibular kinetics: kinesiographic study. Eur J Paediatr Dent. 2008 Mar;9(1):37-42. PMID 18380529
- [Background] Oliveira-Campelo NM, Rubens-Rebelatto J, Marti N-Vallejo FJ, Alburquerque-Sendi N F, Fernandez-de-Las-Penas C. The immediate effects of atlanto-occipital joint manipulation and suboccipital muscle inhibition technique on active mouth opening and pressure pain sensitivity over latent myofascial trigger points in the masticatory muscles. J Orthop Sports Phys Ther. 2010 May;40(5):310-7. doi: 10.2519/jospt.2010.3257. PMID 20436241
- [Background] Cuccia AM, Caradonna C, Annunziata V, Caradonna D. Osteopathic manual therapy versus conventional conservative therapy in the treatment of temporomandibular disorders: a randomized controlled trial. J Bodyw Mov Ther. 2010 Apr;14(2):179-84. doi: 10.1016/j.jbmt.2009.08.002. Epub 2009 Sep 20. PMID 20226365
- [Background] Tuncer AB, Ergun N, Tuncer AH, Karahan S. Effectiveness of manual therapy and home physical therapy in patients with temporomandibular disorders: A randomized controlled trial. J Bodyw Mov Ther. 2013 Jul;17(3):302-8. doi: 10.1016/j.jbmt.2012.10.006. Epub 2012 Nov 16. PMID 23768273
- [Background] Kalamir A, Pollard H, Vitiello A, Bonello R. Intra-oral myofascial therapy for chronic myogenous temporomandibular disorders: a randomized, controlled pilot study. J Man Manip Ther. 2010 Sep;18(3):139-46. doi: 10.1179/106698110X12640740712374. PMID 21886424
- [Background] Kalamir A, Graham PL, Vitiello AL, Bonello R, Pollard H. Intra-oral myofascial therapy versus education and self-care in the treatment of chronic, myogenous temporomandibular disorder: a randomised, clinical trial. Chiropr Man Therap. 2013 Jun 5;21:17. doi: 10.1186/2045-709X-21-17. eCollection 2013. PMID 23738586
- [Background] Guarda-Nardini L, Stecco A, Stecco C, Masiero S, Manfredini D. Myofascial pain of the jaw muscles: comparison of short-term effectiveness of botulinum toxin injections and fascial manipulation technique. Cranio. 2012 Apr;30(2):95-102. doi: 10.1179/crn.2012.014. PMID 22606852
- [Background] Ismail F, Demling A, Hessling K, Fink M, Stiesch-Scholz M. Short-term efficacy of physical therapy compared to splint therapy in treatment of arthrogenous TMD. J Oral Rehabil. 2007 Nov;34(11):807-13. doi: 10.1111/j.1365-2842.2007.01748.x. PMID 17919246
- [Background] Schiffman EL, Look JO, Hodges JS, Swift JQ, Decker KL, Hathaway KM, Templeton RB, Fricton JR. Randomized effectiveness study of four therapeutic strategies for TMJ closed lock. J Dent Res. 2007 Jan;86(1):58-63. doi: 10.1177/154405910708600109. PMID 17189464
- [Background] Nascimento MM, Vasconcelos BC, Porto GG, Ferdinanda G, Nogueira CM, Raimundo RD. Physical therapy and anesthetic blockage for treating temporomandibular disorders: a clinical trial. Med Oral Patol Oral Cir Bucal. 2013 Jan 1;18(1):e81-5. doi: 10.4317/medoral.17491. PMID 23229236
- [Background] Haketa T, Kino K, Sugisaki M, Takaoka M, Ohta T. Randomized clinical trial of treatment for TMJ disc displacement. J Dent Res. 2010 Nov;89(11):1259-63. doi: 10.1177/0022034510378424. Epub 2010 Aug 25. PMID 20739691
- [Background] Shaffer SM, Brismee JM, Sizer PS, Courtney CA. Temporomandibular disorders. Part 2: conservative management. J Man Manip Ther. 2014 Feb;22(1):13-23. doi: 10.1179/2042618613Y.0000000061. PMID 24976744
- [Background] Sterling M, Jull G, Wright A. Cervical mobilisation: concurrent effects on pain, sympathetic nervous system activity and motor activity. Man Ther. 2001 May;6(2):72-81. doi: 10.1054/math.2000.0378. PMID 11414776
- [Background] de Felicio CM, de Oliveira MM, da Silva MA. Effects of orofacial myofunctional therapy on temporomandibular disorders. Cranio. 2010 Oct;28(4):249-59. doi: 10.1179/crn.2010.033. PMID 21032979
- [Background] Mulet M, Decker KL, Look JO, Lenton PA, Schiffman EL. A randomized clinical trial assessing the efficacy of adding 6 x 6 exercises to self-care for the treatment of masticatory myofascial pain. J Orofac Pain. 2007 Fall;21(4):318-28. PMID 18018993
- [Background] La Touche R, Fernandez-de-las-Penas C, Fernandez-Carnero J, Escalante K, Angulo-Diaz-Parreno S, Paris-Alemany A, Cleland JA. The effects of manual therapy and exercise directed at the cervical spine on pain and pressure pain sensitivity in patients with myofascial temporomandibular disorders. J Oral Rehabil. 2009 Sep;36(9):644-52. doi: 10.1111/j.1365-2842.2009.01980.x. Epub 2009 Jul 14. PMID 19627454